CLINICAL TRIAL: NCT03256812
Title: Efficacy and Stability of an Information and Communication Technology (ICT)-Based Centralized Monitoring System for Arrhythmia Detection After Atrial Fibrillation Ablation: a Prospective, Randomized Controlled, Multicenter Study
Brief Title: ICT-based Monitoring for Arrhythmia Detection After AF Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government); Korea Evaluation Institute of Industrial Technology (Other); Daegu Metropolitan City, Korea (Other Government); ICT Clinical Trial Coordination Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ICT_CM_P03_AF
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2019-03

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation
Keywords: Arrhythmias, Atrial Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICT-based ECG monitoring group (Experimental): Continuous monitoring with ICT-based ECG monitoring will begin from the time of participation in the trial in the ICT-based monitoring group. Depending on the lifestyle pattern of the patient, the specific time will be set to allow 30 min of monitoring per day, even if there are no symptoms. If symptoms do appear, additional monitoring will be performed for at least 10 more minutes. 24-hr Holter monitoring will be implemented at the 3-, 6-, and 12-month follow-ups in this group, as in the Holter monitoring group.
  Interventions: Device: ICT-based ECG monitoring
- Holter monitoring group (Active Comparator): 24-hr Holter monitoring will be implemented at the 3-, 6-, and 12-month follow-ups in the Holter monitoring group
  Interventions: Device: Holter monitoring

INTERVENTIONS:
Device: ICT-based ECG monitoring — Continuous monitoring will begin from the time of participation in the trial in the ICT-based centralized monitoring group. 24-hr Holter monitoring will be implemented at the 3-, 6-, and 12-month follow-ups in this group, as in the Holter monitoring group. If heart rate drops below 40 beats/min or increases above 120 beats/min on ECG during ICT-based ECG home monitoring, the participant will be notified first through an alarm function.
  Arms: ICT-based ECG monitoring group
Device: Holter monitoring — 24-hr Holter monitoring will be implemented at the 3-, 6-, and 12-month follow-ups
  Arms: Holter monitoring group

SUMMARY:
To compare the efficacy and stability of an ICT-based centralized clinical trial monitoring system against the efficacy and stability of an existing outpatient-based electrocardiogram (ECG) and Holter monitoring system for arrhythmia detection after atrial fibrillation ablation, and to test whether such continuous monitoring can better detect arrhythmia that is undetectable by existing methods and how this may affect treatment outcomes

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomized, controlled, multicenter study in patients who are capable of using and consent to use a smartphone-based ECG monitoring after ablation for atrial fibrillation. The patients will be randomly assigned to either the Holter monitoring or ICT-based centralized clinical trial monitoring system group in a 1:1 ratio and will undergo monitoring from immediately after the procedure to 12 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years, but < 80 years
2. Patients with non-valvular atrial fibrillation
3. Patients with sustained atrial fibrillation despite ≥ 6 weeks of continuous antiarrhythmia therapy or those who underwent an ablation procedure for tachy-bradycardia syndrome within the previous week
4. Patients who can be followed-up for at least 3 months after ablation
5. Patients who can use and consent to use smartphone-based ECG monitoring
6. Patients who can use a smartphone (Android, version 5.0 or lower; development planned for version 6.0 or higher)
7. Those who can connect to the internet via LAN or WiFi and are in an environment where they can use a gateway and smartphone.

Exclusion Criteria:

1. Patients who cannot be monitored by a smartphone or Bluetooth device
2. Patients who cannot use a smartphone, Bluetooth device, or the internet due to old age
3. Patients with contraindications to standard therapy, such as continued anticoagulant therapy before and after atrial fibrillation ablation
4. Patients belonging to a population vulnerable to clinical trials

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The difference in arrhythmia detection rate | 12 months
  The difference in arrhythmia detection rate between Holter monitoring and ICT-based centralized monitoring

SECONDARY OUTCOMES:
The difference in the number of hospital visits | 12 months
  The difference in the number of hospital visits during the study period due to arrhythmia
The difference in the recurrence rate of atrial fibrillation or atrial tachycardia | 12 months
  The difference in the recurrence rate of atrial fibrillation or atrial tachycardia within 1 year from atrial fibrillation ablation

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Seob Park, MD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea